CLINICAL TRIAL: NCT01472315
Title: Postmenopausal Women,Treatment of Sleep Apnea and Co-morbidities
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1/2000-15
Record Dates: First submitted 2011-10-03; First posted 2011-11-16 (Estimated); Last update posted 2013-03-11 (Estimated); Status verified 2013-03

CONDITIONS: Sleep Apnea
Keywords: sleep apnea; women; postmenopause; hormone treatment
MeSH Terms: conditions — Sleep Apnea Syndromes | interventions — Medroxyprogesterone Acetate

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- medroxyprogesterone acetate (Active Comparator)
  Interventions: Drug: medroxyprogesterone acetate
- Placebo (Placebo Comparator): Placebo pills taken in the same way as the active comparator
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: medroxyprogesterone acetate — MPA hormone therapy 30mg two hours before bedtime and 30mg right before going to bed every night for two weeks period
  Arms: medroxyprogesterone acetate
Drug: Placebo — Placebo pills were taken in same way as active comparator
  Arms: Placebo

SUMMARY:
The purposes of this study are to evaluate the degree and duration of medroxyprogesterone acetate effect as well as tolerability in postmenopausal women with nasal continuous positive airway pressure (CPAP) treated sleep apnea and to compare the effects with nasal CPAP.

DETAILED DESCRIPTION:
Sleep apnea is a common condition affecting both genders. It is affecting more often males than females but after menopause the prevalence of sleep apnea increases in females compared to premenopausal ones and is nearly as high as in males. Continuous positive airway pressure (CPAP) device is the best and standard treatment for the disease. All patients are not adherent to the CPAP treatment and new methods are needed. At the moment no medication is available for sleep apnea. Progesterone hormone is a known respiratory stimulant. Menopause alters significantly women's hormonal balance, for example progesterone levels decrease. Progesterone has been investigated in the treatment of sleep apnea but mostly with male and small populations and the results have been conflicting. Progestins (like medroxyprogesterone acetate, MPA) are female hormones and act through progesterone receptors, so it would be likely women to have less side effects from MPA therapy than men. The purposes of the present study are to evaluate the degree and duration of MPA effect as well as tolerability in postmenopausal women with nasal CPAP treated sleep apnea and to compare the effects with nasal CPAP.

The study is a placebo-controlled double-blind parallel group trial. We included 34 postmenopausal women (17 in placebo and 17 in MPA group) who had been treated for their sleep apnea with CPAP for 1 to 8 years. The trial included measurements at baseline with CPAP, after 14 days of placebo or MPA (60 mg daily) and after three-week washout. The patients discontinued their CPAP one week after the baseline measurements, when they went on with medication. The patients were allowed to continue additional two cycles of MPA treatment before continuing their normal CPAP treatment if they wanted to. Those who continued the additional MPA cycles had the same measurements as in visit 3. The measurements included questionnaires about their symptoms and possible adverse events of MPA, Visual analog scale (VAS) questionnaire with 14 items of sleep quality, Epworth Sleepiness Scale (ESS) and the quality of life questionnaire. Laboratory assays included blood hemoglobin concentration, hematocrit and WBC count, serum creatinine, alanine aminotransferase, total cholesterol, and triglycerides, high-density lipoprotein, estradiol, FSH and thyroid-stimulating hormone and serum MPA concentrations. Overnight polygraphic sleep studies included simultaneous recordings of electroencephalogram (EEG), electro-oculogram (EOG), chin electromyogram (EMG), and electrocardiogram (ECG). Respiration was monitored with a finger probe pulse oximeter (Ohmeda Biox 3700 Pulse Oximeter, BOC Health Care, USA), side-stream capnograph (Datex Normocap® CO2 & O2 Monitor, Instrumentarium, Finland) and the static-charge-sensitive bed (SCSB). During the first visit's CPAP study, Autoset was used in a treatment mode. In the morning after sleep study, subjects completed a questionnaire inquiring their subjective sleep quality during the study night.

ELIGIBILITY:
Inclusion Criteria:

* postmenopausal female
* regular controls of CPAP treatment in pulmonary clinic and regular use of CPAP device

Exclusion Criteria:

* severe or unstable chronic illnesses
* heavy current smoking (over 10 cigarettes per day)
* medication which effects on the central nervous system
* contraindications to progesterone therapy and current participation in any other clinical study

Ages: 42 Years to 77 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2000-01; Primary Completion 2000-11 (Actual); Study Completion 2000-11 (Actual)

PRIMARY OUTCOMES:
polysomnography measures of sleep apnea and sleep | first visit, after 14 days of MPA/placebo use and after 3 weeks washout period
  Sleep stages, apnea-hypopnea index, overnight oxygen saturation values and capnograph values.

SECONDARY OUTCOMES:
subjective questionnaires | first visit, after 14 days of MPA/placebo use and after 3 weeks washout period
  Questionnaires about subjects' symptoms and possible adverse events of MPA, Visual analog scale (VAS) questionnaire with 14 items of sleep quality, Epworth Sleepiness Scale (ESS) and the quality of life questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Sleep Research Unit, Department of Physiology, Turku University, Turku, Finland